CLINICAL TRIAL: NCT04157595
Title: Mackenzie's Mission: The Australian Reproductive Carrier Screening Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); The University of New South Wales (Other); The University of Western Australia (Other); Harry Perkins Institute of Medical Research (Unknown); University of Sydney (Other); Macquarie University, Australia (Other); Griffith University (Other); Victorian Clinical Genetics Services (Unknown); NSW Health Pathology (Unknown); PathWest Laboratory Medicine WA (Other Government); King Edward Memorial Hospital (Other); Royal Brisbane and Women's Hospital (Other Government); Women's and Children's Hospital, Australia (Other Government); Sydney Children's Hospitals Network (Other); Royal Hobart Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RCH HREC 2019.097
Record Dates: First submitted 2019-10-21; First posted 2019-11-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: X-Linked Genetic Diseases; Autosomal Recessive Disorder
Keywords: reproductive genetics; carrier screening; rare disease
MeSH Terms: conditions — Genetic Diseases, X-Linked; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participating Couples (Experimental): Reproductive Genetic Carrier Screening
  Interventions: Other: Reproductive Genetic Carrier Screening

INTERVENTIONS:
Other: Reproductive Genetic Carrier Screening — Carrier screening for approximately 1300 genes associated with severe autosomal recessive and X-linked recessive conditions affecting children will be performed on each member of the couple. A combined result will be issued indicating whether the couple has a 'low' or 'increased' risk of having a child with a genetic condition

SUMMARY:
This study will investigate reproductive genetic carrier screening (RGCS) in 10,000 couples across Australia. Carrier screening for approximately 1300 genes associated with severe, childhood-onset, X-linked and autosomal recessive conditions will be performed on each member of the couple. A combined result will be issued indicating whether the couple has a 'low' or 'increased' risk of having a child with a genetic condition. It is anticipated that 1-2% of couples will be at an increased risk of having an affected child.

The study will evaluate all aspects of the RGCS program to assess the feasibility and acceptability of a publicly-funded population-wide RGCS program, including:

* education of recruiting healthcare providers
* education of participating couples
* implementation and uptake of RGCS
* frequency of increased-risk couples and their reproductive decisions
* psychosocial impacts
* ethical issues
* health economic implications
* health implementation research

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

Couples will be invited to take part in the study by their healthcare provider (HCP). The couple will enrol via an online portal, complete an education module, provide consent and complete a questionnaire. Those who consent to carrier screening will be sent mouth swab kits with samples returned by mail.The carrier screening performed will be done via accredited testing laboratories in partnership with clinical genetics services. Genetic counselling will be available to study participants throughout the process. Couples at increased risk will be offered a genetic counselling consultation and offered support to access reproductive options (i.e. prenatal diagnosis, preimplantation genetic diagnosis (PGD) which will be funded by the study for one cycle of IVF with PGD). All participants will be asked to complete an initial survey at study enrolment and invited to complete optional surveys at the time of screening, after return of screening results, and approximately 13 to 19 months after results. Subsets of participants will also be invited to take part in interviews.

GENE LIST FOR CARRIER SCREENING

The approximately 1300 genes tested in the Mackenzie's Mission carrier screening panel meet the following criteria:

1. The associated condition is one where an 'average' couple would take steps to prevent the birth of a child with that condition.

   - This includes conditions with significant negative impact on quality of life for the child, the condition being lethal in childhood, and a significant impact on the family.
2. AND/OR: There is a potential benefit for knowing about the condition to inform management in the neonatal period. This criterion was particularly important if the condition was either not included on a newborn screening panel, and/or intervention would be required prior to results from newborn screening being known.
3. AND there is strong evidence for mutations in the gene being causative of the condition in question, with enough variants reported to allow confidence in informing couples of their chance of having a child with the condition in question.

ELIGIBILITY:
In order to take part in the study, couples need to have visited a recruiting HCP who will assess them for eligibility based on the criteria below:

INCLUSION CRITERIA

* Planning to become pregnant or in early pregnancy (less than 10 weeks gestation at enrolment and less than 11 weeks gestation at sample receipt by the laboratory)
* Both members of the couple available to participate in the study and available to provide a sample for testing at the same time.
* If the couples are using an egg/sperm donor/s, the donor/s need to be available to provide a DNA sample for testing and consent to having carrier screening.

NB: If both members of the couple are known carriers of the same autosomal recessive condition, or the female is a known carrier of an X-linked recessive condition, they will still be eligible to have RGCS through the study, but will only be considered an 'increased-risk' couple for the purposes of this study if they are identified through the study testing to be carriers of pathogenic variants in a different gene.

EXCLUSION CRITERIA

Participating couples meeting any of the following requirements will be excluded from this study:

* Pregnant and greater than 10 weeks gestation at enrolment.
* Only one member of the couple agrees to participate in the study.
* One or both members of the couple are less than 18 years old.
* Both members of the couple are not available to be tested at the same time.
* The couple are using an egg/sperm donor/s and the donor/s are not available for testing or the couple are using an anonymous donor.
* One member of the couple has already been screened as part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18302 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Screening Uptake (Quantitative) | At offer of screening
  Practitioners offering screening will be asked to record the number of couples offered screening which will allow calculation of screening uptake.
Frequency of Increased-Risk Couples | At reporting of results (~Weeks 5-6 since enrolment)
  Analysis of carrier frequencies of the genes tested and the frequency of identification of increased-risk couples
Reproductive Choices made by Increased-Risk Couples | Reproductive choices made by couples will be tracked from the date an increased-risk result is received until study closure on 31 December 2022. A subset of couples will be interviewed ~19 months after receiving an increased-risk result.
  For pregnant couples, the investigators will ascertain how many have prenatal diagnosis (PND), and of those who have PND and an affected fetus is identified, how many terminate the pregnancy. For those who are not pregnant at the time of screening, the investigators will ascertain choices for future pregnancies that occur during the timeframe of the study, including how many choose preimplantation genetic diagnosis (PGD), how many choose a naturally conceived pregnancy with PND and how many choose a naturally conceived pregnancy without any testing.
Cohort Characteristics of those who decline and those who accept RGCS | Couples who decline screening;at offer or at enrolment (Day 0); optional. Couples who accept screening; at enrolment (Day 0); compulsory.
  Short survey capturing personal information: age, country of birth, language spoken at home, ethnicity, religion and religiosity, education level, employment status, household income, marital status, pregnancy history and family/genetic history information.
Predictors of Uptake - Decliners | Couples who decline screening; at offer or enrolment (Day 0); optional
  Survey asking main reason(s) for declining to participate informed by the Health Belief Model (HBM). The HBM is used to predict and explain uptake of a health behaviour. It includes four components: perceived benefits, perceived susceptibility, perceived severity and perceived barriers (Janz and Becker 1984). A subset of declining couples will be invited for interview to explore the decision-making process and their reasons for declining testing.
Predictors of Uptake - Decliners | At decision not to provide samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  Survey asking main reason(s) for declining to participate informed by the Health Belief Model (HBM). The HBM is used to predict and explain uptake of a health behaviour. It includes four components: perceived benefits, perceived susceptibility, perceived severity and perceived barriers (Janz and Becker 1984). A subset of declining couples will be invited for interview to explore the decision-making process and their reasons for declining testing.
Predictors of Uptake - Acceptors | Couples who accept screening; at offer or enrolment (Day 0); compulsory.
  Survey asking main reason(s) for choosing to participate informed by the Health Belief Model (HBM). The HBM is used to predict and explain uptake of a health behaviour. It includes four components: perceived benefits, perceived susceptibility, perceived severity and perceived barriers (Janz and Becker 1984)
Predictors of Uptake - Acceptors | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  Survey asking main reason(s) for choosing to participate informed by the Health Belief Model (HBM). The HBM is used to predict and explain uptake of a health behaviour. It includes four components: perceived benefits, perceived susceptibility, perceived severity and perceived barriers (Janz and Becker 1984)

SECONDARY OUTCOMES:
Participant Experience - Attitudes/Perceptions | Couples who decline screening;at offer or at enrolment (Day 0); optional. Couples who accept screening; at enrolment (Day 0); compulsory.
  Survey assessing attitudes towards carrier screening in the general population, and the attitudes of the couple towards carrier screening for themselves.
Participant Experience - State-Anxiety - pre-screening | Couples who decline screening; at enrolment (Day 0); optional. Couples who accept screening; at enrolment (Day 0); compulsory.
  Six-item short-form of the state-anxiety scale of the Spielberger State-Trait Anxiety Inventory (STAI) (Marteau and Bekker 1992). This scale measures how the respondent feels "right now, at this moment". Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - State-Anxiety - pre-screening II | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  Six-item short-form of the state-anxiety scale of the Spielberger State-Trait Anxiety Inventory (STAI) (Marteau and Bekker 1992). This scale measures how the respondent feels "right now, at this moment". Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - State-Anxiety - post-result | Low-risk and increased-risk couples; post-result (~Weeks 17-18 since enrolment); optional
  Six-item short-form of the state-anxiety scale of the Spielberger State-Trait Anxiety Inventory (STAI) (Marteau and Bekker 1992). This scale measures how the respondent feels "right now, at this moment". Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - State-Anxiety - long-term follow-up | Low-risk couples; long-term follow-up (~13 months since enrolment); optional. Increased-risk couples; long-term follow-up (~19 months since enrolment); optional
  Six-item short-form of the state-anxiety scale of the Spielberger State-Trait Anxiety Inventory (STAI) (Marteau and Bekker 1992). This scale measures how the respondent feels "right now, at this moment". Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - Trait-Anxiety - pre-screening | Couples who decline screening; at enrolment (Day 0); optional. Couples who accept screening; at enrolment (Day 0); compulsory.
  20-item trait-anxiety scale (Form Y2) of the Spielberger State-Trait Anxiety Inventory (STAI). This scale measures how the respondent "generally" feels. Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - Trait-Anxiety - pre-screening II | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  20-item trait-anxiety scale (Form Y2) of the Spielberger State-Trait Anxiety Inventory (STAI). This scale measures how the respondent "generally" feels. Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - Trait-Anxiety - post-result | Low-risk and increased-risk couples; post-result (~Weeks 17-18 since enrolment); optional
  20-item trait-anxiety scale (Form Y2) of the Spielberger State-Trait Anxiety Inventory (STAI). This scale measures how the respondent "generally" feels. Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Participant Experience - Trait-Anxiety - long-term follow-up | Low-risk couples; long-term follow-up (~13 months since enrolment); optional. Increased-risk couples; long-term follow-up (~19 months since enrolment); optional
  20-item trait-anxiety scale (Form Y2) of the Spielberger State-Trait Anxiety Inventory (STAI). This scale measures how the respondent "generally" feels. Scores range from 20 to 80. A high score indicates the presence of high levels of anxiety.
Health Economic Impact - Assessment of Quality of Life - pre-screening | Couples who decline testing, at enrolment (Day 0); optional. Couples who accept testing, at enrolment (Day 0); compulsory
  12-item Assessment of Quality of Life-4D (AQoL-4D) questionnaire (Hawthorne, Richardson and Osbourne 1999; Richardson and Hawthorne 1998). This questionnaire measures health-related quality of life in four dimensions: Independent Living, Relationships, Mental Health and Senses. Total scores range from a minimum of 12 to a maximum of 48. Higher scores indicate a lower health-related quality of life.
Health Economic Impact - Assessment of Quality of Life - post-result | Low-risk and increased-risk couples; post-result (~Weeks 17-18 since enrolment); optional
  12-item Assessment of Quality of Life-4D (AQoL-4D) questionnaire (Hawthorne, Richardson and Osbourne 1999; Richardson and Hawthorne 1998). This questionnaire measures health-related quality of life in four dimensions: Independent Living, Relationships, Mental Health and Senses. Total scores range from a minimum of 12 to a maximum of 48. Higher scores indicate a lower health-related quality of life.
Health Economic Impact - Assessment of Quality of Life - long-term follow-up | Low-risk couples; long-term follow-up (~13 months since enrolment); optional. Increased-risk couples; long-term follow-up (~19 months since enrolment); optional
  12-item Assessment of Quality of Life-4D (AQoL-4D) questionnaire (Hawthorne, Richardson and Osbourne 1999; Richardson and Hawthorne 1998). This questionnaire measures health-related quality of life in four dimensions: Independent Living, Relationships, Mental Health and Senses. Total scores range from a minimum of 12 to a maximum of 48. Higher scores indicate a lower health-related quality of life.
Health Economic Impact - Participants' willingness to pay | Couples who decline screening, at enrolment (Day 0); optional. Couples who accept screening, at enrolment (Day 0); compulsory
  Questions with randomised monetary values to assess maximum amount participants would be willing to pay, and whether the test should be government, privately or Medicare funded.
Participant Experience - Health Literacy | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  Questions to assess health literacy level
Participant Experience - Evaluation of Educational and Decision-Aid Materials | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  Questions to evaluate resources developed for participating couples e.g. decision aid, website, brochure
Participant Experience - Decisional Conflict | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  16-item scale measuring personal perception of uncertainty, factors contributing to uncertainty, and effective decision making. Includes five subscores: uncertainty, informed, values clarity, support, effective decision making (O'Conner 1993 (updated 2010)). Total scores range from 0 [no decisional conflict] to 100 [very high decisional conflict].
Participant Experience - Deliberation | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  6-item scale measuring decision deliberation. Dichotomous scale: responses below the midpoint (11 or under) classified as not deliberated and those at or above the midpoint as deliberated (Van den Berg, Timmermans, Ten et al 2006)
Participant Experience - Decision-Making Approach | At provision of samples for screening, anticipated to be within ten days of enrolment (Days 2-10); optional
  Survey evaluating decision-making approach i.e. whether it was an individual or shared decision and who was involved in the decision-making process, e.g. couples, family, health-professional
Participant Experience - Genomics Outcome Scale (GOS-6) | Increased-risk couples, before and after genetic counselling session (~Weeks 5-6 since enrolment)
  6-item scale measuring empowerment as an outcome of clinical genetics services. Total scores range from a minimum of 6 to a maximum of 30. Higher scores indicate higher levels of empowerment (Grant et al. 2018)
Participant Experience - Decisional Regret - post-result | Low-risk and increased-risk couples; post-result (~Weeks 17-18 since enrolment); optional
  A 5-item scale measuring distress and remorse after a health care decision. Scores range from 0 [no regret] to 100 [high regret]. Subset of low-risk couples to be contacted for interview to explore experience of having testing and receiving a low-risk result.
Participant Experience - Decisional Regret - long-term follow-up | Low-risk couples; long-term follow-up (~13 months since enrolment); optional. Increased-risk couples; long-term follow-up (~19 months since enrolment); optional
  A 5-item scale measuring distress and remorse after a health care decision. Scores range from 0 [no regret] to 100 [high regret]. Subset of low-risk couples to be contacted for interview to explore experience of having testing and receiving a low-risk result.
Participant Experience - Qualitative Interviews | Low-risk couples; long-term follow-up (~13 months since enrolment); optional. Increased-risk couples; long-term follow-up (~19 months since enrolment); optional
  Subset of low-risk couples to be contacted for interview to explore longer-term experience of having testing and receiving a low-risk result. Subset of increased-risk couples to be contacted for interview to explore the experience of receiving a increased-risk result, the use of this information in reproductive decision-making, and the communication of genetic information within families.

OTHER OUTCOMES:
Ethical Issues - Assessment of ethical aspects of publicly funded preconception screening | Throughout study; 3 years
  A series of scholarly outputs (e.g. journal articles) critically considering ethical issues in publicly funded preconception screening programs. The issues being identified include (but are not limited to) reproductive autonomy, public health ethics frameworks, eugenics, secondary findings. Additional ethical issues will be considered as they arise in the trial. The method to be used is applied ethics, which is non-empirical.
Implementation Outcomes - Barriers & Enablers to Implementation | Study investigators; at committee meetings for the duration of the study (3 years); Jan 2019 - Dec 2022
  Barriers and enablers to implementation will be identified and recorded at study committee meetings via responses to the following questions: What has changed over the last month or so? What has gone well/not so well? Has anything surprised you?
Implementation Outcomes - Anticipated vs Actual Outcomes | Study investigators; 1 month before the study begins recruitment
  To assess whether planned and anticipated outcomes are realised, study investigators will be asked to complete a time-capsule survey predicting the outcomes of the study. Following the completion of the study, the responses will be matched to the final outcomes.
Implementation Outcomes - Patient Safety Behaviour Questionnaire | HCPs; at HCP conferences or professional meetings; for the duration of the study (3 years).
  Questionnaire assessing what HCPs in the wider community think about carrier screening, and what the barriers/enablers are to offering carrier screening to patients in usual care.
Implementation Outcomes - Uptake by HCPs | HCPs; at invitation to become a recruiting HCP; for the duration of the study (3 years)
  Survey of HCPs invited to recruit to the study, including those who agree to recruit couples and those who decline to recruit couples. The survey will explore potential barriers to RGCS, factors that might influence confidence/ability to refer appropriate couples for RGCS and readiness to change. HCPs can opt-in to be contacted for interview to provide further information about implementation.
Implementation Outcomes - Factors influencing Recruitment by HCPs - post-education | Recruiting HCPs; 3 months after education
  Survey of HCPs who agree to recruit to the study, measuring factors influencing recruitment such as knowledge, ability and confidence.
Implementation Outcomes - Factors influencing Recruitment by HCPs - post-recruitment | Recruiting HCPs; 6 weeks after recruitment of first participant
  Survey of HCPs who have recruited to the study, measuring factors influencing recruitment. Opt-in to be contacted for interview to further explore the experience of offering RGCS to patients and any barriers/enablers of implementation.
Implementation Outcomes - HCP Experience - post-implementation | Recruiting HCPs; 3 months after end of recruitment
  Survey of HCPs who have recruited to the study, examining their experience of offering reproductive genetic carrier screening.
Health Economic Impact - Costs per increased-risk couple identified | 3 months after enrolment
  Cost in Australian dollars of identifying one increased-risk couple
Health Economic Impact - Costs per affected pregnancy identified | 6 months after enrolment
  Cost in Australian dollars of identifying one affected pregnancy
Health Economic Impact - Costs per affected birth averted | Throughout study; 3 years
  Average cost in Australian dollars of taking reproductive measures to avoid having an affected live birth (e.g. pre-implantation genetic diagnosis, prenatal diagnosis, termination etc.)
Health Economic Impact - Costs of the carrier screening program | Throughout study; 3 years
  Total costs of the carrier screening program

CONTACTS AND LOCATIONS:
Overall Officials: Martin Delatycki, Principal Investigator — Murdoch Children's Research Institute/Victorian Clinical Genetics Services; Edwin Kirk, Principal Investigator — Sydney Children's Hospital Network/NSW Health Pathology/UNSW; Nigel Laing, Principal Investigator — University of WA/Harry Perkins Institute/PathWest Laboratory Medicine
Locations (24):
- Australia (24):
  - Forster Community Health Service, Forster, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Hunter Genetics, Newcastle, New South Wales
  - Royal Hospital for Women, Sydney, New South Wales
  - Sydney Children's Hospital, Randwick, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Campbelltown Hospital, Sydney, New South Wales
  - Tamworth Communith Health Services, Tamworth, New South Wales
  - Taree Community Health Service, Taree, New South Wales
  - Wagga Wagga Base Hospital, Wagga Wagga, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Mareeba Hospital, Mareeba, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Victorian Clinical Genetics Services, Melbourne, Victoria
  - Northern Hospital, Melbourne, Victoria
  - Mercy Hospital for Women, Melbourne, Victoria
  - West Gippsland Heath Service (Warragul Hospital), Warragul, Victoria
  - Joondalup Health Campus, Joondalup, Western Australia
  - King Edward Memorial Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified samples, genomic data and associated clinical information may be shared with researchers for other Human Research Ethics Committee approved research studies and with recognised national and international databases to advance scientific knowledge.

REFERENCES:
- [Derived] Kirk EP, Delatycki MB, Archibald AD, Tutty E, Caruana J, Halliday JL, Lewis S, McClaren BJ, Newson AJ, Dive L, Best S, Long JC, Braithwaite J, Downes MJ, Scuffham PA, Massie J, Barlow-Stewart K, Kulkarni A, Ruscigno A, Kanga-Parabia A, Rodrigues B, Bennetts BH, Ebzery C, Hunt C, Cliffe CC, Lee C, Azmanov D, King EA, Madelli EO, Zhang F, Ho G, Danos I, Liebelt J, Fletcher J, Kennedy J, Beilby J, Emery JD, McGaughran J, Marum JE, Scarff K, Fisk K, Harrison K, Boggs K, Giameos L, Fitzgerald L, Thomas L, Burnett L, Freeman L, Harris M, Berbic M, Davis MR, Cifuentes Ochoa M, Wallis M, Wall M, Chow MTM, Ferrie MM, Pachter N, Quayum N, Lang N, Kasi Pandy P, Casella R, Allcock RJN, Ong R, Edwards S, Sundercombe S, Jelenich S, Righetti S, Lunke S, Kaur S, Stock-Myer S, Eggers S, Walker SP, Theodorou T, Catchpool T, Clinch T, Roscioli T, Hardy T, Zhu Y, Fehlberg Z, Boughtwood TF, Laing NG; Mackenzie's Mission Investigators; Mackenzie's Mission Investigators. Nationwide, Couple-Based Genetic Carrier Screening. N Engl J Med. 2024 Nov 21;391(20):1877-1889. doi: 10.1056/NEJMoa2314768. PMID 39565987